CLINICAL TRIAL: NCT03617692
Title: Effects of Cannabis Use in Cancer Patients: A Feasibility Study
Brief Title: Cannabis Use in Cancer Patients
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 18-0836.cc
Record Dates: First submitted 2018-07-23; First posted 2018-08-06 (Actual); Results first posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Solid Tumor, Adult
Keywords: Cannabis; Tumors; Observational Study
MeSH Terms: conditions — Marijuana Abuse; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Oral Cannabis: This is an observational study of individuals who have already decided to try cannabis for their cancer treatment-related symptoms. A research assistant will provide information on the range of edible cannabis products and basic information about their various cannabinoid profiles, approximate prices, and nearby locations where participants may choose to purchase their product. Participants will then initiate use of an orally administered product they have selected and obtained. Participants will take the product as they see fit, without any frequency or dosing instructions from study staff, for two weeks.

SUMMARY:
The goal of this study is to determine the feasibility of a human observational study of orally administered cannabis use among cancer patients.

DETAILED DESCRIPTION:
Tightly controlled experimental laboratory studies (e.g., clinical trials with randomization) using Cannabis products available in state-regulated markets are simply, at this point, not possible owing largely to federal law and the University requirements related to the Controlled Substances Act and Drug Free Schools and Communities Act. Because a traditional clinical trial design is not possible given the current federal status of Cannabis products, this investigator will use a patient-oriented, prospective observational design. Specifically, individuals who have already decided to try Cannabis for their cancer treatment-related symptoms will initiate use of an orally administered product they have selected. A research assistant will provide information on the range of edible cannabis products and basic information about their various cannabinoid profiles, approximate prices, and nearby locations where participants may choose to purchase their product. The participants will then purchase the product and decide how often and how much to use. This approach is consistent with federal law and supported by our preliminary and ongoing studies(1R01AT009541-01, 1R01DA044131-01, CDPHE2902, R01DA039707). Patients will take the product as they see fit, without any frequency or dosing instructions from study staff, for two weeks, at which time they will be scheduled for an acute administration session (Ta1-Tc1) so that we may examine the acute effects of the product. The final follow-up will be one month later via an online survey sent directly to the participant via email.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Provision to sign and date the consent form.
2. Stated willingness to comply with all study procedures and be available for the duration of the study.
3. Be a female or male aged at least 21 years.
4. Have a diagnosis of any solid tumor type who has or is undergoing either curative or palliative treatment
5. Have intent or interest to use cannabis to treat their symptoms.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Report of other non-prescription drug use, such as cocaine, heroin, methamphetamine in the past 60 days
2. Actively seeking or in treatment for any substance use disorder
3. Acute illness other than cancer that could affect cognition or compliance per the decision of the study M.D.
4. Premenopausal females who are pregnant or trying to become pregnant. Note that pregnancy testing will not be required.
5. A Telephone Interview for Cognitive Status (TICS) score indicating moderate or severe cognitive impairment at screening

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or females, ages 21 and up, with a diagnosis of any solid tumor type who has or is undergoing either curative or palliative treatment
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Bryan, PhD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado Hospital, Aurora, Colorado
  - University of Colorado Boulder, Boulder, Colorado

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oral Cannabis
Started | 27
Completed | 24
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Oral Cannabis
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 22
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Likelihood of Accruing Participants: Feasibility of Enrollment
Description: Enroll a minimum of 30 patients and demonstrate reasonable compliance with study procedures within 54 months of active recruiting.
Time Frame: Approximately 48 months
Population: Number of participants assessed for enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Cannabis
Number analyzed (Participants) | 41
Participants
  Enrolled | 27
  Completed study | 24

2. Other Pre Specified Outcome: Amount of Interest
Description: Study officials will document how many patients contact the research team regarding their participation in the study
Time Frame: Approximately 48 months
Population: Number of individuals who contacted the research team about participation in the study
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Cannabis
Number analyzed (Participants) | 134
Participants | 134

3. Other Pre Specified Outcome: Eligibility
Description: Study officials will document how many patients are and are not eligible to participate in the study.
Time Frame: Approximately 48 months
Population: Number of individuals who contacted the research team about participation in the study
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Cannabis
Number analyzed (Participants) | 134
Participants
  Eligible after pre-screening | 41
  Not eligible after pre-screening | 5
  Did not complete pre-screening | 88

4. Other Pre Specified Outcome: Enrollment
Description: Study officials will document how many patients actually proceed to enrollment in the study.
Time Frame: Approximately 48 months
Population: Number of individuals found eligible after pre-screening
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Cannabis
Number analyzed (Participants) | 41
Participants
  Enrolled | 27
  Not enrolled | 14

5. Other Pre Specified Outcome: Completion of Assessments
Description: Study officials will document how many participants complete each assessment (baseline assessment, pre-acute cannabis use assessment, 1 hour post-acute cannabis use, 2 hour post-acute cannabis use, one month follow up assessment).
Time Frame: Baseline to one month follow up, Approximately 48 months
Population: Number of participants enrolled
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Cannabis
Number analyzed (Participants) | 27
Participants
  Completed baseline assessment | 27
  Completed pre-acute cannabis use assessment | 25
  Completed 1 hour post-acute cannabis use assessment | 25
  Completed 2 hour post-acute cannabis use assessment | 25
  Completed one month follow up assessment | 24

6. Other Pre Specified Outcome: Study Completion
Description: Study officials will document how many participants complete the study in its entirety.
Time Frame: Approximately 48 months
Population: Number of participants enrolled
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Cannabis
Number analyzed (Participants) | 27
Participants | 24

ADVERSE EVENTS:
Time Frame: 3 months
Description: Participants were asked about the occurrence of adverse events at study visits.
Arm/Group | Oral Cannabis
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 1/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Cannabis (N=27)
Increased heart rate (over 100 beats per minute) (Cardiac disorders) | 1 (1) — Heart rate observed to be over 100 beats per minute during a study visit

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-31): https://cdn.clinicaltrials.gov/large-docs/92/NCT03617692/Prot_SAP_000.pdf